CLINICAL TRIAL: NCT02594215
Title: Phase 1 Dose Finding Trial of MK-7075 in Children and Adults With Proteus Syndrome
Brief Title: Dose Finding Trial of MK-7075 in Children and Adults With Proteus Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 160014; 16-HG-0014
Record Dates: First submitted 2015-10-31; First posted 2015-11-03 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Proteus Syndrome
Keywords: AKT1; Overgrowth
MeSH Terms: conditions — Proteus Syndrome | interventions — Miransertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Experimental
  Interventions: Drug: MK-7075 (miransertib)

INTERVENTIONS:
Drug: MK-7075 (miransertib) — MK-7075 or miransertib (formerly ARQ 092) is small molecule that effectively inhibits AKT. Proteus syndrome is caused by mosaic activating mutations in AKT1. This is a phase I study to determine a recommended dose for subsequent trials, which will determine the efficacy of miransertib in Proteus syndrome.

SUMMARY:
Background:

Proteus syndrome (PS) is caused by a mutation in the AKT1 gene. This gene makes a protein that communicates with other proteins in the body to make cells grow. The AKT1 mutation changes chemical signals in the body and causes overgrowth. PS can be fatal. The drug MK-7075 reduces signals from the AKT1 protein. This may reduce or stabilize some of the overgrowth in people with PS. Researchers want to find the best dose of MK-7075 based on its effect on tissues in people with PS.

Objective:

To determine the safety, tolerability, and recommended dose of MK-7075 in people with PS.

Eligibility:

People ages 6 and older with PS

Design:

Participants will be screened with medical history, physical exam, and blood and urine tests.

Participants will take MK-7075 by mouth once daily for up to 12 28-day cycles.

Participants must stay near the NIH Clinical Center (CC) during the whole first cycle, for weekly visits to the CC. For cycle 2, they will have visits every 2 weeks. They will have 1 visit before cycles 3 and 4, and once before every other cycle for cycles 5 11. The final visit will be at the end of cycle 12. Visits may include:

Small skin samples taken.

ECG: Soft electrodes on the skin record heart signals.

Echocardiogram: A small probe held to the chest takes pictures of the heart.

MRI: Participants will lie in a machine that takes pictures of the body.

Joint and mobility function tests.

Participants will complete surveys by phone and in person.

Participants will keep a daily medication and symptom diary.

...

DETAILED DESCRIPTION:
Proteus syndrome is a rare segmental overgrowth disorder caused by a somatic gain of function mutation, c.49GA, p.Glu17Lys) in the oncogene AKT1, encoding the AKT1 kinase . The disorder is progressive, with high morbidity and mortality - there are very few living adults with this disease. Tissues and cell lines from patients with Proteus syndrome harbor admixtures of mutant alleles that ranged from <1% to approximately 50%. This mutation causes constitutive activation of AKT1, through Ser473 and Thr308 phosphorylation. This activation stimulates the AKT/PI3K pathway, mediating processes including increased cell proliferation and decreased apoptosis. The progressive nature of the disorder and the mechanism of disease (gain of function) make AKT1 an excellent target for therapeutics, specifically repression. The AKT/PI3K pathway is mutated in numerous cancers as well. Because it is commonly mutated in cancer, pharmaceutical companies are interested in targeting this molecule with inhibitors. Indeed, Proteus syndrome can be considered a simple model for cancer therapeutics, as these patients are known to harbor only a single activating mutation instead of the hundreds or thousands that are mutated in cancers. ArQule Inc., a wholly owned subsidiary of Merck & Co., has developed a small molecule, miransertib (MK-7075) that effectively inhibits AKT, with the lowest IC50 for AKT1 (as compared to AKT2 or AKT3, and orders of magnitude lower for other kinases). This agent has undergone significant development with animal toxicity studies and is currently in phase I trials in patients with different types of cancer. In addition, we have performed in vitro testing with miransertib in cells from patients with Proteus syndrome and demonstrated reduction in AKT1 phosphorylation at doses in the range of achievable blood levels in humans with low toxicity. Because Proteus syndrome is a chronic disease, typical approaches to defining the recommended phase II dose by determining the maximum tolerated dose (MTD) are not appropriate it is unreasonable to propose that patients would tolerate significant side effects for prolonged time periods. As an initial trial for this disease, we propose a phase I study to determine a recommended dose for subsequent trials, which will determine the efficacy of miransertib in Proteus syndrome. The recommended phase II dose will be determined based on the tolerability of miransertib in children and adults with Proteus syndrome and measures of drug levels in plasma and affected tissues in patients with Proteus syndrome and measures of tissue phosphorylation of AKT1. We hypothesize that the recommended dose of miransertib will be substantially below that of doses used in patients with cancer and that this will lead to a highly favorable risk-benefit ratio on which we can base future efficacy studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Meets published clinical criteria for PS.
* Measurable disease: Patients must have at least one measurable lesion for volumetric MRI or photographic CCTN.
* Has a CLIA-validated report demonstrating presence of a mosaic AKT1 c.49G>A mutation.
* 6 years of age or older. The age limits including children and adolescents were chosen because childhood and puberty are considered to be the greatest risk for disease progression, and MK-7075 may provide the most benefit to this young group of patients. In addition, an important objective of this study is to characterize the pharmacokinetics of MK-7075 in the pediatric population since it has been better studied in adults.
* Not using nor has used within the past 6 months any medication known to affect the AKT/PI3K pathway (e.g., everolimus), reviewed by NIHCC pharmacist.
* Performance status: Patients greater than or equal to 16 years of age must have a Karnofsky performance level of greater than or equal to 40%, and adolescents 6 - 16 years old must have a Lansky performance of greater than or equal to 40%.
* Is willing to identify and allow us to communicate with an outside medical provider if needed.
* Hepatic function: Bilirubin must be less than or equal to 1.5 x the upper limit of normal and the SGPT (ALT) must be less than or equal to 2.5 x the upper limit of normal.
* Cardiac function: Must have an ejection fraction with normal limits for age by echocardiogram.
* Must have cognitive abilities to complete patient surveys/QOL assessments as appropriate for age or have an appropriate surrogate decision-maker or guardian able to complete these measures in the case of intellectually impaired adults.
* Renal function: Age-adjusted normal serum creatinine (see Table below) OR a creatinine clearance greater than or equal to 60 mL/min/1.73 m^2.

  * Age (Years): less than or equal to 15; Serum Creatinine (mg/dl): less than or equal to1.2
  * Age (Years): > 15; Serum Creatinine (mg/dl): less than or equal to 1.5
* Body surface area of at least 0.5 m^2

EXCLUSION CRITERIA:

* Pregnant or breast-feeding females are excluded due to potential risks of fetal and teratogenic adverse events of an investigational agent. Pregnancy tests must be obtained prior to enrollment on this study in all females. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. Abstinence is an acceptable method of birth control.
* Patients who anticipate the need for surgical intervention within the first three cycles (3 months), as surgical intervention during the period of DLT evaluation may affect analysis of adherence and/or make the subject unevaluable.
* An investigational agent within the past 6 months.
* Ongoing radiation therapy, chemotherapy, hormonal therapy directed at the disease, immunotherapy, or biologic therapy.
* Clinically significant unrelated systemic illness, such as serious infections, hepatic, renal or other organ dysfunction, which in the judgment of the Principal or Associate Investigator would compromise the patient s ability to tolerate the agents used in this trial or are likely to interfere with the study procedures or results.
* Type I or II diabetes mellitus or is being treated with insulin or an oral hypoglycemic agent.
* Abnormal LVEF on echocardiogram.
* Patients with known extensive intestinal involvement of the disease or evidence of malabsorption that, in the investigator s opinion could compromise drug absorption.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Inability to undergo MRI/CT and/or contraindication for MRI examinations following the MRI protocol. Prosthesis or orthopedic or dental braces that would interfere with volumetric analysis of target lesion on MRI.
* Evidence of a tumor, or other cancer requiring treatment with chemotherapy or radiation therapy.
* Patients with baseline (pre-treatment) QTcF>470ms on ECG.
* Absence of an approved legal guardian or approved surrogate decision-maker in the case of intellectually impaired adults.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Tissue drug levels | End of cycle 3
  Tissue drug levels are assessed at baseline, cycle 1 /day 14, and cycle 4/day 1.
Tissue phospho-AKT level | End of cycle 3
  Tissue tissue phospho-AKT is assessed at baseline, cycle 1/day 14, and cycle 4/day 1.
Tolerabilty/Side Effects | Ongoing
  Tolerability and side effects are assessed on an ongoing basis.

SECONDARY OUTCOMES:
Tolerability and side effects | Ongoing
  Tolerability and side effects are assessed on an ongoing basis.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie G Biesecker, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Ours CA, Sapp JC, Hodges MB, de Moya AJ, Biesecker LG. Case report: five-year experience of AKT inhibition with miransertib (MK-7075) in an individual with Proteus syndrome. Cold Spring Harb Mol Case Stud. 2021 Dec 9;7(6):a006134. doi: 10.1101/mcs.a006134. Print 2021 Dec. PMID 34649967
- [Derived] Keppler-Noreuil KM, Sapp JC, Lindhurst MJ, Darling TN, Burton-Akright J, Bagheri M, Dombi E, Gruber A, Jarosinski PF, Martin S, Nathan N, Paul SM, Savage RE, Wolters PL, Schwartz B, Widemann BC, Biesecker LG. Pharmacodynamic Study of Miransertib in Individuals with Proteus Syndrome. Am J Hum Genet. 2019 Mar 7;104(3):484-491. doi: 10.1016/j.ajhg.2019.01.015. Epub 2019 Feb 22. PMID 30803705
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-HG-0014.html